CLINICAL TRIAL: NCT04364308
Title: The Relationship Between Umbilical Cord ph and Feto-maternal Doppler Studies in Scheduled Nonlaboring Term Singleton Caesarean Deliveries
Status: Suspended | Type: Observational
Why Stopped: No found.
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, MD, research , gynecology and obstetrics, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 358
Record Dates: First submitted 2020-04-19; First posted 2020-04-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Fetal Hypoxia; Fetal Conditions
Keywords: Fetal Doppler; Ultrasound exam; cesarean delivery; umbilical cord ph; scheduled cesarean delivery; cerebroplacental ratio
MeSH Terms: conditions — Fetal Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fetal Echography — Fetal ultrasound and its parameters

SUMMARY:
Perinatal asphyxia is a crucial reason for neonatal and childhood morbidity and death. Fetal and neonatal acidemia can be utilised as predictors for establishing such risk. Several researches have reported a marked relation between low values of fetal pH with short- and long-term adverse neonatal outcomes. Umbilical cord blood gas studies (UCGS) are considered critical data that gives an objective and certified evaluation of the oxygenation and metabolic status of the fetus. Before birth, the physician can evaluate fetal wellness through cardiotocography and prenatal ultrasound. Other studies had examined the role of fetal Doppler indices before birth and proposed that fetuses with lower impedance in the middle cerebral artery (MCA) or low cerebroplacental ratio (CPR) are at increased risk of adverse pregnancy outcome. However, no research has ever evaluated the possibility of a correlation between ultrasonographic fetal evaluation and fetal umbilical cord pH as a predictor of pre-delivery fetal pH.

The goal of our study was to discovered a potential association between the venous umbilical ph cord blood at delivery and the ultrasonographic feto-maternal doppler indices in patients with a scheduled nonlaboring term singleton caesarean deliveries (SCD), this research is a novel finding.

DETAILED DESCRIPTION:
the investigators included in our study only singleton term (37 0/7 - 41 6/7 weeks of gestation) pregnancies delivered by a scheduled nonlaboring term singleton caesarean deliveries.

This was an observational study carried out at a single university tertiary care center

For every patient, an ultrasound examination was performed within one day of delivery and the fetal doppler indices were recorded. The umbilical venous pH were obtained immediately after delivery and before placental detachment with heparinized syringes

The primary endpoints were CPR, umbilical (UA) and fetal MCA arteries indices. The second endpoints analysed when measurable were ductus venosus (DV) and uterine artery (Ut) pulsatility indices, all indices were examined using colour Doppler ultrasound according to a standard procedure and CPR was evaluated as the ratio between the MCA and UA pulsatility indices.

The venous umbilical cord pH at birth was correlated with ultrasound doppler parameters, calculating the correlation coefficient r2 and P-value. Statistical significance was fixed at P<0.05. the investigators performed a linear regression analysis to find the association between the different ultrasound indices and the venous pH.

ELIGIBILITY:
Inclusion Criteria:

* singleton term (37 0/7 - 41 6/7 weeks of gestation) pregnancies delivered by a scheduled nonlaboring term singleton caesarean deliveries

Exclusion Criteria:

* Pregnancies complicated by fetal malformations, stillbirth, preterm deliveries.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the investigators enrolled only pregnant women
Study Population: the investigators enrolled only low-risk pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The venous umbilical cord pH at birth was correlated with ultrasound doppler parameters | pre-intervention
  the investigators recordered venous umbilical cord pH and all fetal doppler parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi della Campania "Luigi Vanvitelli"- OB & Gyn -, Napoli, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided